CLINICAL TRIAL: NCT03491540
Title: Mechanical Bowel Preparation and Oral Antibiotics Before Rectal Cancer Surgery: a Multi Center Double-Blinded Randomized Controlled Trial (PREPACOL2 Study)
Brief Title: Mechanical Bowel Preparation and Oral Antibiotics Before Rectal Cancer Surgery
Acronym: PREPACOL2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P160938J
Record Dates: First submitted 2018-03-09; First posted 2018-04-09 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Rectal Cancer Surgery
Keywords: Mechanical Bowel Preparation (MBP); Oral antibiotics; Rectal cancer surgery; Surgical site infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Gentamicins; Ornidazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both participants and investigators are unaware of the intervention assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1) " MBP and oral antibiotics " group (Experimental): Sennosides colonic preparation Oral Gentamycin Oral Ornidazole
  Interventions: Drug: Sennosides colonic preparation; Drug: Oral Gentamycin; Drug: Oral Ornidazole
- 2) " MBP alone " group (Placebo Comparator): Sennosides colonic preparation Oral placebo Gentamycin Oral placebo Ornidazole
  Interventions: Drug: Sennosides colonic preparation; Drug: Oral Placebo Gentamycin; Drug: Oral Placebo Ornidazole

INTERVENTIONS:
Drug: Sennosides colonic preparation — Mechanical bowel preparation :
  Sennosides colonic preparation (X-PREP)
  1 per day, on day -2 and day -1
Drug: Oral Gentamycin — Oral gentamycin:
  Gentamycin 80 mg, 4 per day, on day -2 and day -1; Liquid forms in individual vials
  Arms: 1) " MBP and oral antibiotics " group
Drug: Oral Ornidazole — Oral ornidazole :
  Ornidazole
  1 g per day (2 tablet per day), on day -2 and day -1; In tablets
  Arms: 1) " MBP and oral antibiotics " group
Drug: Oral Placebo Gentamycin — Placebo for oral gentamycin :
  Same presentation as oral gentamycin x4 per day on day -2 and day -1
  Arms: 2) " MBP alone " group
Drug: Oral Placebo Ornidazole — Placebo for oral ornidazole :
  Same presentation as oral ornidazole
  1g per day (2 tablets per day) on day -2 and day -1
  Arms: 2) " MBP alone " group

SUMMARY:
This study aims to demonstrate that a preoperative combination of mechanical bowel preparation and oral antibiotics, before elective laparoscopic rectal cancer surgery, is associated with a reduction of postoperative surgical site infection rate, as compared to mechanical bowel preparation alone Our hypothesis is that a preoperative colonic preparation including a combination of mechanical bowel preparation and oral antibiotics before elective laparoscopic rectal cancer surgery is associated with a reduced rate of 30-day postoperative surgical site infection, as compared to mechanical bowel preparation alone

DETAILED DESCRIPTION:
This study aims to demonstrate that a preoperative combination of mechanical bowel preparation and oral antibiotics, before elective laparoscopic rectal cancer surgery, is associated with a reduction of postoperative surgical site infection rate, as compared to mechanical bowel preparation alone.

This study's hypothesis is that a preoperative colonic preparation including a combination of mechanical bowel preparation and oral antibiotics before elective laparoscopic rectal cancer surgery is associated with a reduced rate of 30-day postoperative surgical site infection, as compared to mechanical bowel preparation alone Preoperative mechanical bowel preparation (MBP) has been proposed in an attempt to reduce the colonic fecal load and to limit the risk of surgical site contamination, thus theoretically limiting the risk of postoperative surgical site infection (SSI). However, the benefit of such MBP before colorectal surgery is related to type of procedure performed. Indeed, several randomized controlled trials (RCT) and meta-analyses have demonstrated the absence of benefit of MBP before colon cancer surgery, whereas a recent RCT suggested that MBP before rectal cancer surgery was associated to a significant reduction of postoperative SSI, as compare to the absence of preoperative MBP.

Recent studies suggested that the adjunction of oral antibiotics during MBP could help efficiently reduce the risk of postoperative SSI. Indeed, a recent meta-analysis of RCT have suggested that patients preoperatively receiving both MBP and oral antibiotics were exposed to a significantly reduced risk of postoperative SSI, as compared to patients receiving only preoperative MBP. This result was confirmed in a recent RCT which compared preoperative MBP and oral antibiotics versus MBP alone in a heterogeneous population of patients who underwent laparoscopic colonic or rectal surgery. However, to date, no RCT compared the outcomes of an MBP with oral antibiotics to MBP without oral antibiotics in a homogeneous cohort of patients undergoing rectal cancer surgery.

This study aims to demonstrate that a preoperative combination of mechanical bowel preparation and oral antibiotics, before elective laparoscopic rectal cancer surgery, is associated with a reduction of postoperative surgical site infection rate, as compared to mechanical bowel preparation alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or more
* Scheduled to undergo elective restorative laparoscopic cancer of the rectal (<15 cm from the anal margin) with sphincter preservation
* With Signed consent
* And affiliated to the French social security system

Exclusion Criteria:

* Emergent surgery
* Scheduled total colo-proctectomy
* Scheduled abdominoperineal restion with definitive colostomy
* Scheduled associated concomitant resection of another organ (liver, etc.)
* Active bacterial infection at the time of surgery or recent antibiotic therapy (up to 15 days before surgery)
* Associated inflammatory bowel disease
* Patients with known colonization with multidrug-resistant enterobacteriacea
* History of allergy or contraindication to the Ornidazole, Gentamycin, X-PREP or to any of the excipients of the drugs used.
* Cirrhosis of grade B and C (Child-Pugh classification)
* Myasthenia
* Allergy to one of the other treatments administered for the purpose of the trial (including betadine)
* Patient suffering from severe central neurologic diseases, fixed or progressive.
* Pregnant patients
* Refusal to participate or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Postoperative 30-day surgical site infection (SSI). | 30 days
  SSI will be defined and classified as superficial, deep and/or organ-space infection on the basis of validated and well-defined criteria developed by the Centers for Disease Control and Prevention (CDC), validated in French by the Comité technique des infections nosocomiales et des infections liées aux soins.

SECONDARY OUTCOMES:
Overall postoperative morbidity | 30 days
  Including all postoperative complications occurring within 30 days after surgery, defined and classified according to the Clavien-Dindo classification.
Severe postoperative morbidity | 30 days
  Including all complications graded 3 or more according to the Clavien-Dindo classification, and occurring within 30 days after surgery.
Postoperative mortality | 30 days
  Including all deaths occurring within 30 days after surgery.
Postoperative anastomotic leakage | 90 days
  Defined as the passing of any intra-colonic content (air, liquid, intestinal content, or radiological contrast) through an anastomosis or by an peri-anastomotic abscess, even in the absence of intra-colonic content leak through the anastomosis, observed in drainages, surgical incision, vagina, during a surgical procedure or on a radiological examination, occurring within 90 days after surgery.
Postoperative length of hospital stay | Up to 90 days
  Calculated from the day of surgery to the day of hospital discharge.
Unplanned hospitalization | 90 days
  Defined as any unplanned hospitalization between surgery and postoperative day 90.
Tolerance of the colonic preparation | The day before surgery
  Evaluated using a dedicated questionnaire performed the evening before surgery.
Clostridium difficile colitis occurrence | 30 days
  Defined as clinical symptoms of clostridium difficile colitis with at least 1 stool sample positive for Clostridium difficile toxin A/B as detected by enzyme-linked immunosorbent assay within 30 days after surgery.
Rate of multi-resistant bacteria carriage | The day before or the day of surgery
  Defined as rate of multi-resistant bacteria carriage
Date of adjuvant chemotherapy beginning | 90 days
  If indicated
Temporary stoma closure rate | 90 days
  Define as temporary stoma closure

CONTACTS AND LOCATIONS:
Locations (1):
- Service de chirurgie viscérale, cancérologique / Hôpital Saint-Louis, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] Willis MA, Toews I, Soltau SL, Kalff JC, Meerpohl JJ, Vilz TO. Preoperative combined mechanical and oral antibiotic bowel preparation for preventing complications in elective colorectal surgery. Cochrane Database Syst Rev. 2023 Feb 7;2(2):CD014909. doi: 10.1002/14651858.CD014909.pub2. PMID 36748942